CLINICAL TRIAL: NCT07248592
Title: Empathy Training: Its Effect on Maternity Nurses' Communication and Parturient Women's Perception of Empathetic Care
Brief Title: Empathy Training and Its Effect on Maternity Nurses' Communication Skills
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Nadia Youssef Ahmed AbdElla, assistant professor, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 0593
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Communication Skills; Patient Satisfaction
Keywords: Maternity nurses; empathetic communication skills; women perception; Parturient women
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: This study employs a single-group pre-test/post-test design. One cohort of maternity nurses will receive the intervention. Outcomes are measured at baseline (pre-test) before the training begins and then again after the training is complete (post-test). The primary analysis will compare the outcomes from these two time points to assess the effect of the training.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Empathy and Communication Skills Training Arm (Experimental): This arm consists of all enrolled study participants, who are qualified maternity nurses working in the labor and delivery unit at Mansoura University Hospitals .
  Interventions: Other: Maternity Nurse Empathy and Communication Skills Training Program

INTERVENTIONS:
Other: Maternity Nurse Empathy and Communication Skills Training Program — All participants in this single arm will receive the structured MNECS Training Program. This is a multi-session, interactive workshop designed to enhance empathy and patient-centered communication.
  Other Names: MNECS Training Program

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of empathy skills training on Maternity Nurses' Communication and Parturient Women's Perception of Empathetic Care.

The main questions it aims to answer are;

* Do maternity nurses who received empathy skills training have better empathetic communication skills when caring with parturient women than those who don't.?
* Do parturient women who received care from maternity nurses trained with empathy skills training perceive higher empathy level than mothers who received care from untrained nurses?

Participants will:

* Have 3 educational training sessions on empathy communication skills.
* Will be followed by the researcher for any clarifications about the educational content of session
* nurses will be asked to evaluate their empathy communication skills twice (once before training and second time after training) .

also parturient women will be asked to assess their maternity nurses' empathy care level twice (once before training and second time after training).

DETAILED DESCRIPTION:
Empathy is one of the elements that influence compassionate skills which required for building a meaningful relationship between maternity nurse and the patient requires. Empathy is particularly important to maternity nurse and allows them to understand things from a woman's angle. Indeed, nurses with high-empathy are able to comprehend the feelings of women, which are very beneficial, particularly during some stages of childbirth when women may not want to talk or in situations where verbal communication is not possible. However, providing effective and empathic communication between maternity nurse and mothers increases satisfaction and control over delivery and reduces blood pressure, anxiety, pain, and fear of childbirth.

This study used a quasi-experimental (one group pre/posttest) . it will be conducted at three health settings at Mansoura city, Egypt and will involve 45 maternity nurses and 120 parturient women. Maternity nurses will be trained on empathic communication skills.

ELIGIBILITY:
Inclusion Criteria:

* Be currently employed in a maternity care setting Labor & Delivery Unit.
* Have direct patient contact with parturient women as a primary part of their regular duties.
* Have a minimum of 6 months of experience.

Exclusion Criteria:

* Nurses whose primary role is administrative, managerial without direct patient care responsibilities.
* Have previously participated in a pilot or feasibility study for the same or a highly similar intervention.
* Planned absence (e.g., extended leave, vacation) for a significant portion of the study intervention or data collection period.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Maternity Nurses' Empathy and Communication skills | one week after ending sessions of training
  Empathy level among maternity nurses, measured using the Toronto Empathy Questionnaire (TEQ). The total score ranges from 0 to 64, with a higher score indicating greater empathy.

SECONDARY OUTCOMES:
Parturient Women Perception of Maternity Nurses' Empathic Care | one week after ending sessions of training
  Parturient women's perception of nurses' empathic care, measured using the Consultation and Relational Empathy (CARE) Measure. The total score ranges from 10 to 50, with a higher score indicating better perceived empathy.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Y AbdElla, Assis. prof, Principal Investigator — Mansoura University
Locations (1):
- Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
The reason for not sharing data is to comply with and protect the confidentiality of participants, which is a primary ethical requirement in research.